CLINICAL TRIAL: NCT00609518
Title: Pemetrexed With Simplified Folate and Dexamethasone Supplementation Versus Pemetrexed With Standard Supplementation as Second-line Chemotherapy for Patients With Non-squamous Non-small Cell Lung Cancer
Brief Title: A Study for Patients With Non-Squamous Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Chief Medical Officer, Eli Lilly
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 11652; H3E-CR-S111 (Other: Eli Lilly and Company)
Record Dates: First submitted 2008-01-23; First posted 2008-02-07 (Estimated); Results first posted 2010-11-15 (Estimated); Last update posted 2010-12-28 (Estimated); Status verified 2010-12

CONDITIONS: Non Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Pemetrexed; Folic Acid; Vitamin B 12; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard Vitamin and Steroid Schedule + Pemetrexed (Active Comparator): Standard vitamin and steroid schedule that is used with pemetrexed consisting of a minimum of 5 daily doses of folic acid before first pemetrexed dose and dexamethasone on day before, day of, and day after treatment.
  Interventions: Drug: pemetrexed; Dietary Supplement: Folic acid; Dietary Supplement: Vitamin B12; Drug: dexamethasone
- Simplified Vitamin and Steroid Schedule + Pemetrexed (Experimental): Simplified vitamin and steroid schedule to be used with pemetrexed consisting of 2 daily doses of folic acid before first pemetrexed dose and dexamethasone on day of treatment only.
  Interventions: Drug: pemetrexed; Dietary Supplement: Folic Acid; Dietary Supplement: Vitamin B12; Drug: dexamethasone

INTERVENTIONS:
Drug: pemetrexed — 500 mg/m^2 intravenous infusion on day 1 of each 21-day cycle. Number of Cycles: Until progression or to a maximum of 6 cycles.
  Other Names: Alimta; LY231514
Dietary Supplement: Folic acid — 350-1000 micrograms taken orally for at least 5 daily doses during the 7-day period prior to the first dose of pemetrexed then continues daily throughout treatment until 3 weeks after the last dose of pemetrexed.
  Other Names: Folate
  Arms: Standard Vitamin and Steroid Schedule + Pemetrexed
Dietary Supplement: Folic Acid — 350-1000 micrograms taken orally for two consecutive daily doses of folic acid the day before and the day of the first dose of pemetrexed the continues throughout treatment and for 3 weeks after the last dose of pemetrexed.
  Other Names: Folate
  Arms: Simplified Vitamin and Steroid Schedule + Pemetrexed
Dietary Supplement: Vitamin B12 — 1000 micrograms intramuscular injection of vitamin B12 during the week prior to the first dose of pemetrexed then further injections given approximately every 9 weeks until 3 weeks after the last dose of pemetrexed.
Drug: dexamethasone — 4 mg taken orally [or equivalent] twice per day the day before, the day of, and the day after the first day of pemetrexed. Continue to give dexamethasone twice per day the day before, the day of, and the day after each dose of pemetrexed.
  Arms: Standard Vitamin and Steroid Schedule + Pemetrexed
Drug: dexamethasone — 4 mg taken orally [or equivalent] twice per day on the day of the first dose of pemetrexed. Continue to give dexamethasone twice per day on the day of each dose of pemetrexed.
  Arms: Simplified Vitamin and Steroid Schedule + Pemetrexed

SUMMARY:
Chemotherapy for patients with non-squamous non-small cell lung cancer. Patients are given folic acid, vitamin B12 and steroids, both before and during treatment, to reduce the side effects associated with pemetrexed. The aim is whether it is possible to simplify the folic acid and steroid schedule without increasing toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Histologic or cytologic diagnosis of non-small cell lung cancer (NSCLC) with locally advanced or metastatic disease (Stage IIIA, IIIB or IV)that is of non-squamous histology
* Patients must have failed only one prior chemotherapy regime and must be considered eligible for further chemotherapy following progression of their disease.
* Eastern Cooperative Oncology Group (ECOG) performance status 0 to 2
* Adequate organ function

Exclusion Criteria:

* Concurrent administration of any other anti-tumor therapy
* Other co-existing malignancies
* Pregnancy or breast feeding
* Serious concomitant disorders
* Inability or unwillingness to take folic acid or vitamin B12 supplementation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 111 (Actual)
Dates: Start 2008-02; Primary Completion 2009-10 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (14):
- Australia (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bankstown, New South Wales
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Concord, New South Wales
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kingswood Penrith, New South Wales
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Liverpool, New South Wales
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Redcliffe, Queensland
- Italy (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bologna
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Milan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Napoli
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Pisa
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Rome
- Mexico (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mexico City
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Toluca
- Spain (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Pozuelo de Alarcón
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Seville

REFERENCES:
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Completed is defined as:The patient has completed follow-up visits until 12 months after the randomization date.
  Qualified Intent-to-Treat (Q-ITT) is defined as: Include all randomized patients, with nonsquamous histology, who comply with their pretreatment folic acid and steroid supplementation schedule and take at least one dose of pemetrexed.
Period: Overall Study
Arm/Group | Standard Vitamin and Steroid Schedule + Pemetrexed | Simplified Vitamin and Steroid Schedule + Pemetrexed
Started | 54 | 57
Completed 6 Treatment Cycles | 19 | 22
Completed | 11 | 17
Not Completed | 43 | 40
Not completed — Death from Study Disease | 32 | 32
Not completed — Withdrawal by Subject | 5 | 3
Not completed — Lost to Follow-up | 3 | 0
Not completed — Physician Decision | 1 | 3
Not completed — Death from Adverse Event | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Vitamin and Steroid Schedule + Pemetrexed | Simplified Vitamin and Steroid Schedule + Pemetrexed | Total
Number analyzed (Participants) | 54 | 57 | 111
Age Continuous [Mean (Standard Deviation); unit: years] | 62.1 (11.08) | 60.9 (12.13) | 61.4 (11.60)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 18 | 40
  Male | 32 | 39 | 71
Region of Enrollment [Number; unit: participants]
  Spain | 8 | 9 | 17
  Mexico | 27 | 27 | 54
  Italy | 15 | 18 | 33
  Australia | 4 | 3 | 7
Eastern Cooperative Oncology Group (ECOG) Performance Status [Number; unit: participants] — Classifies patients according to their functional impairment. Scores range from 0 (Fully Active) to 5 (Death).
  participants
    0- Fully Active | 26 | 26 | 52
    1- Ambulatory, Restricted Strenuous Activity | 28 | 28 | 56
    2- Ambulatory, No Work Activities | 0 | 2 | 2
    Not Assessed | 0 | 1 | 1
Smoking Status [Number; unit: Participants]
  Past Smoker | 32 | 33 | 65
  Never Smoked | 14 | 15 | 29
  Current Smoker | 8 | 9 | 17
Pathological Diagnosis [Number; unit: Participants]
  Cytological | 17 | 21 | 38
  Histopathological | 37 | 36 | 73
Disease Stage [Number; unit: Participants] — Stage means how big the tumor is and how far it has spread. Stages range from 0 (not spread) to IV (spread throughout the body). Differentiation between stage IIIA and IIIB is in accordance with the American Joint Committee on Cancer Staging Criteria for Lung Cancer.
  Participants
    IIIA | 3 | 1 | 4
    IIIB | 9 | 13 | 22
    IV | 42 | 43 | 85
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] — Body mass index is an estimate of body fat based on body weight divided by height squared (kilograms/square meters [kg/m^2]).
  kg/m^2 | 25.3 (3.98) | 26.0 (5.20) | 25.7 (4.64)

OUTCOME MEASURES:

1. Primary Outcome: Safety: Number of Participants With Drug-Related Grade 3 or 4 Toxicity
Description: Results are presented for the number of participants with drug-related Grade 3 or 4 toxicity/adverse event (AE). Grades range from 0 (none) to 5 (death), with Grade 3 and 4 being defined as follows:
  Grade 0 = No AE; Grade 1 = Mild AE; Grade 2 = Moderate AE; Grade 3 = Severe AE; Grade 4 = Life-threatening or disabling AE; Grade 5 = Death related to AE. A detailed list of Serious and non-serious adverse events is provided in the Reported Adverse Event section.
Time Frame: From first dose of treatment to last dose of treatment plus 30 days
Population: Qualified Intention to Treat (Q-ITT)
Measure: Number; unit: participants
Arm/Group | Standard Vitamin and Steroid Schedule + Pemetrexed | Simplified Vitamin and Steroid Schedule + Pemetrexed
Number analyzed (Participants) | 51 | 47
participants | 15 | 18
Statistical Analysis 1: Comparison: Standard Vitamin and Steroid Schedule + Pemetrexed vs Simplified Vitamin and Steroid Schedule + Pemetrexed; Test type: Superiority or Other; Linear probability model; Risk Difference (RD) = 0.09, 95% CI 2-sided [-0.10 to 0.28]

2. Secondary Outcome: Proportion of Participants With Best Overall Tumor Response (Response Rate)
Description: Response defined per Response Evaluation Criteria In Solid Tumors (RECIST) criteria: Complete Response (CR)=disappearance of all target lesions; Partial Response (PR)=30% decrease in sum of longest diameter of target lesions; Progressive Disease=20% increase in sum of longest diameter of target lesions; Stable Disease=small changes that do not meet above criteria. Best Overall Tumor Response is complete response plus partial response.
Time Frame: Baseline until disease progression, new therapy initiated, or death from any cause, up to 12 months after enrollment.
Population: Qualified Intent to Treat (Q-ITT)
Measure: Mean (95% Confidence Interval); unit: proportion of patients
Arm/Group | Standard Vitamin and Steroid Schedule + Pemetrexed | Simplified Vitamin and Steroid Schedule + Pemetrexed
Number analyzed (Participants) | 51 | 47
proportion of patients | 0.118 [0.044 to 0.239] | 0.064 [0.013 to 0.175]
Statistical Analysis 1: Comparison: Standard Vitamin and Steroid Schedule + Pemetrexed vs Simplified Vitamin and Steroid Schedule + Pemetrexed; Test type: Superiority or Other; p = 0.4902, Fisher Exact

3. Secondary Outcome: Overall Survival
Description: Overall survival is the duration from randomization to death. For patients who are alive, overall survival is censored at the date of last contact.
Time Frame: Randomization (≤4 weeks from baseline visit) to 12 months after randomization
Population: Qualified Intent to Treat (Q-ITT)
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Standard Vitamin and Steroid Schedule + Pemetrexed | Simplified Vitamin and Steroid Schedule + Pemetrexed
Number analyzed (Participants) | 51 | 47
months | 8.2 [5.4 to 11.7] | 9.2 [7.6 to 11.3]
Statistical Analysis 1: Comparison: Standard Vitamin and Steroid Schedule + Pemetrexed vs Simplified Vitamin and Steroid Schedule + Pemetrexed; Test type: Superiority or Other; p = 0.6791, Log Rank
Statistical Analysis 2: Comparison: Standard Vitamin and Steroid Schedule + Pemetrexed vs Simplified Vitamin and Steroid Schedule + Pemetrexed; Test type: Superiority or Other; Regression, Cox; Treatment was the covariate included in this model; Hazard Ratio (HR) = 0.90, 95% CI 2-sided [0.54 to 1.49]

4. Secondary Outcome: Progression-free Survival (PFS)
Description: Defined as the time from date of first dose to the first observation of disease progression, or death due to any cause. For patients who are alive and have not progressed, PFS is censored at the date of last radiological assessment.
Time Frame: Randomization (≤4 weeks from baseline visit) to 12 months after randomization
Population: Qualified Intent to Treat (Q-ITT)
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Standard Vitamin and Steroid Schedule + Pemetrexed | Simplified Vitamin and Steroid Schedule + Pemetrexed
Number analyzed (Participants) | 51 | 47
months | 3.7 [2.9 to 4.9] | 3.8 [1.8 to 5.9]
Statistical Analysis 1: Comparison: Standard Vitamin and Steroid Schedule + Pemetrexed vs Simplified Vitamin and Steroid Schedule + Pemetrexed; Test type: Superiority or Other; p = 0.5870, Log Rank
Statistical Analysis 2: Comparison: Standard Vitamin and Steroid Schedule + Pemetrexed vs Simplified Vitamin and Steroid Schedule + Pemetrexed; Test type: Superiority or Other; Regression, Cox; Treatment was the covariate included in this model; Hazard Ratio (HR) = 0.89, 95% CI 2-sided [0.57 to 1.38]

ADVERSE EVENTS:
Arm/Group | Standard Vitamin and Steroid Schedule + Pemetrexed | Simplified Vitamin and Steroid Schedule + Pemetrexed
Serious Adverse Events (participants affected / at risk) | 18/54 | 18/57
Other Adverse Events (participants affected / at risk) | 47/54 | 54/57
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard Vitamin and Steroid Schedule + Pemetrexed (N=54) | Simplified Vitamin and Steroid Schedule + Pemetrexed (N=57)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Pancytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (2) | 0 (0)
Gastrointestinal inflammation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Chest pain (General disorders) | 0 (0) | 2 (2)
Oedema peripheral (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1)
Bronchiectasis (Infections and infestations) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Lobar pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 2 (2) | 1 (1)
Respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Humerus fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Ataxia (Nervous system disorders) | 0 (0) | 1 (1)
Complex regional pain syndrome (Nervous system disorders) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 1 (1) | 1 (1)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
Hydropneumothorax (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Laryngeal oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Oesophagobronchial fistula (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Swelling face (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard Vitamin and Steroid Schedule + Pemetrexed (N=54) | Simplified Vitamin and Steroid Schedule + Pemetrexed (N=57)
Anaemia (Blood and lymphatic system disorders) | 13 (17) | 18 (24)
Leukopenia (Blood and lymphatic system disorders) | 8 (13) | 18 (36)
Lymphopenia (Blood and lymphatic system disorders) | 9 (9) | 15 (20)
Neutropenia (Blood and lymphatic system disorders) | 13 (21) | 17 (31)
Thrombocytopenia (Blood and lymphatic system disorders) | 7 (9) | 7 (8)
Abdominal pain (Gastrointestinal disorders) | 3 (3) | 2 (2)
Constipation (Gastrointestinal disorders) | 3 (3) | 4 (4)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 4 (5)
Nausea (Gastrointestinal disorders) | 11 (15) | 19 (21)
Vomiting (Gastrointestinal disorders) | 6 (10) | 8 (8)
Asthenia (General disorders) | 14 (16) | 14 (14)
Chest pain (General disorders) | 4 (4) | 2 (2)
Fatigue (General disorders) | 6 (7) | 7 (9)
Pyrexia (General disorders) | 0 (0) | 6 (9)
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 (0) | 3 (3)
Alanine aminotransferase increased (Investigations) | 6 (10) | 9 (15)
Aspartate aminotransferase increased (Investigations) | 2 (4) | 6 (11)
Blood alkaline phosphatase increased (Investigations) | 3 (3) | 5 (7)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 3 (3)
Decreased appetite (Metabolism and nutrition disorders) | 1 (2) | 8 (8)
Hyperglycaemia (Metabolism and nutrition disorders) | 4 (4) | 6 (7)
Hyponatraemia (Metabolism and nutrition disorders) | 4 (5) | 8 (9)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3)
Headache (Nervous system disorders) | 3 (3) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 8 (9) | 11 (13)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 7 (8) | 11 (13)
Rash (Skin and subcutaneous tissue disorders) | 8 (8) | 7 (9)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days